CLINICAL TRIAL: NCT03477656
Title: Evaluation of 2 Techniques of Apheresis to Desensitize ABO Incompatible Kidney Transplant Candidates: Double Filtration PlasmaPheresis (DFPP) vs Large Plasma Volume Specific ImmunoAdsorption
Brief Title: Evaluation of 2 Techniques of Apheresis to Desensitize ABO Incompatible Kidney Transplant Candidates
Acronym: DADI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/16/8767
Record Dates: First submitted 2018-02-09; First posted 2018-03-26 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Kidney Transplantation
Keywords: ABO incompatible kidney transplantation; Desensitization; Double Filtration PlasmaPherisis (DFPP); Specific immunoadsorption; Living donor kidney transplantation
MeSH Terms: interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large volume specific immunoadsorption (Experimental): 1 to 2 sessions of large volume specific immunoadsorption according to the initial isoagglutinin titer.
  Interventions: Procedure: Large volume specific immunoadsorption
- Double Filtration Plasmapheresis (Experimental): 1 to 5 sessions of double filtration plasmapheresis according to the initial isoagglutinin titer.
  Interventions: Procedure: Double Filtration Plasmapheresis

INTERVENTIONS:
Procedure: Large volume specific immunoadsorption — 1 to 2 sessions of large volume specific immunoadsorption using GLYCOSORB®-ABO column
  Arms: Large volume specific immunoadsorption
Procedure: Double Filtration Plasmapheresis — 1 to 5 sessions of double filtration plasmapheresis
  Arms: Double Filtration Plasmapheresis

SUMMARY:
Kidney transplantation is the treatment of choice for end-stage renal disease. ABO incompatible (ABOi) living donor kidney transplantation is one of the best ways to expand the donors' pool. However, breaking the ABO barrier is possible only with a preconditioning regimen that includes 1) an immunosuppressive strategy using a B-cell depleting agent (rituximab), an induction therapy with polyclonal antibodies, and a maintenance triple immunosuppressive therapy based on calcineurin inhibitors, and 2) a desensitization protocol aiming to decrease the titer of isoagglutinins. For this purpose, several techniques of apheresis are available. To date, two main techniques used in clinical setting are the Double-Filtration PlasmaPheresis (DFPP) and the Antigen-Specific Immunoadsorption (SIA). DFPP permits the depletion of the selective plasma fraction containing Immunoglobulins, while limiting the need for plasma substitution. SIA enables to remove ABO antibodies without a major loss in essential plasma components. To date, no randomized study comparing DFPP and SIA exist. SIA is less often used because of its high cost. However, in order to reduce the number of SIA sessions and consequently its cost, large plasma volume sessions of SIA are performed. ABOi is dramatically more expensive than ABO compatible kidney transplantation. A large part of the difference in the cost is related to the apheresis technique.

Herein, the investigator proposes to describe the efficacy, the safety, and the cost of DFPP and SIA to desensitize ABO incompatible kidney transplant candidates.

DETAILED DESCRIPTION:
All recipients will receive an induction therapy with rituximab and polyclonal antibodies, as well as a maintenance therapy by tacrolimus, mycophenolic acid (switched for mTOR (Mechanistic target of rapamycin) inhibitors 1 month after the transplantation to avoid viral infections) and steroids.

The desensitization protocol will be based on the initial titer of isoagglutinin. All patients with an isoagglutinin titer between 1/8 and 1/128 will be included in this monocentric, open label study, and randomized between the DFPP arm (1 to 4 sessions according to the initial titer) and large-plasma SIA (1 to 2 sessions according to the titer). The effectiveness will be evaluated on the ability to obtain the targeted titer before transplantation (1/4) with less than 5 DFPP, or 2 large-plasma volume SIA.

All recipients will be followed for 6 months, and examined for surgical complications, rejection rate, and kidney function. All complications related to desensitization protocol will be reported. Moreover, all cost associated with these two apheresis techniques will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for living donor ABO incompatible kidney transplantation
* Presenting an IsoAgglutinin immunoglobulin G titer (anti-A-B) between 1/8 and 1/128, before desensitization
* Patient older than 18 years
* Women of childbearing age must have a pregnancy test before starting the study and undergoing study. They must take an effective and acceptable method of contraception before starting the study and throughout the study period. Sexually active men should use a condom throughout the course of the study
* Patient able to sign an informed consent form
* Patient affiliated with a social security scheme

Exclusion Criteria:

* Presence of anti-HLA (Human Leucocyte Antigens) allo-antibodies
* Patient with comorbidities that prevent desensitization protocols
* Women who are pregnant, or who may become pregnant or breastfeeding women
* History of hypersensitivity related to a component of the apheresis membrane
* Subjects under legal protection
* Subjects participating in another interventional research protocol or in an exclusion period from another interventional research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Success rate | the day of transplantation
  % of subjects with the targeted isoagglutinin titer (≤1/4) before transplantation with less than 5 DFPP sessions (for the DFPP arm) or 2 large plasma volume specific immunoadsorption sessions (for the specific immunoadsorption arm)

SECONDARY OUTCOMES:
Differential cost-efficacy ratio of support for patients receiving a live donor kidney transplant Incompatible ABO and benefiting from a desensitization procedure | 7 months
  Direct medical costs ( treatments costs, costs of hospital stays, costs of outpatient cares) will be evaluated from the society point of view.
  A cost-efficacy analysis, comparative of medical consequences, measured in terms of number of complications related to the technique and post surgical at 7 months, and the economic consequences will be realized.
Surgical complication rate during the desensitization sessions | From the first desensitization session to the last one, assessed up to 10 days
  % of subjects with surgical complications during the desensitization sessions
Surgical complication rate during the transplantation surgery | During the transplantation surgery
  % of subjects with surgical complications during the transplantation surgery
Thrombotic complication rate during the desensitization sessions | From the first desensitization session to the last one, assessed up to 10 days
  % of subjects with thrombotic complications during the desensitization sessions
Thrombotic complication rate 1 week after transplantation surgery | 1 week after transplantation surgery
  % of subjects with thrombotic complications until 1 week after transplantation surgery
Rate of bleeding and/or hematoma on vascular access during the desensitization sessions | From the first desensitization session to the last one, assessed up to 10 days
  % of subjects with bleeding and/or hematoma on vascular access during the desensitization sessions
Rate of hematoma occurrence during the transplantation surgery | During the transplantation surgery
  % of subjects with hematoma during the transplantation surgery
Rate of occurrences of hemorrhage away from vascular access during the desensitization sessions | From the first desensitization session to the last one, assessed up to 10 days
  % of subjects with hemorrhage away from vascular access during the desensitization sessions
Rate of occurrences of allergy to the components of the membrane or of the blood circuit (tube set) during the desensitization sessions | From the first desensitization session to the last one, assessed up to 10 days
  % of subjects with allergy to the components of the membrane or of the blood circuit (tube set) during the desensitization sessions
Rate of occurrences of allergy to the components of the membrane or of the blood circuit (tube set) 1 week after transplantation surgery | 1 week after transplantation surgery
  % of subjects with allergy to the components of the membrane or of the blood circuit (tube set) until 1 week after transplantation surgery
Blood transfusion rate before transplantation | Before transplantation
  % of subjects who received blood transfusion before transplantation
Blood transfusion rate during the transplantation surgery | During the transplantation surgery
  % of subjects who received blood transfusion during the transplantation surgery
Blood transfusion rate 1 week after transplantation surgery | 1 week after transplantation surgery
  % of subjects who received blood transfusion until 1 week after transplantation surgery
Occurrence rate of deep vein or graft vein thrombosis during the transplantation surgery | During the transplantation surgery
  % of subjects with deep vein or graft vein thrombosis during the transplantation surgery
Graft ablation rate 1 week after transplantation surgery | 1 week after transplantation surgery
  % of subjects with graft ablation until 1 week after transplantation surgery
Complication rate on surgical area 1 week after transplantation surgery | 1 week after transplantation surgery
  % of subjects with complication on the surgical area until 1 week after transplantation surgery
Infectious complication rate 1 week after transplantation surgery | 1 week after transplantation surgery
  % of subjects with Infectious complication until 1 week after transplantation surgery
Need for dialysis session(s) 1 week after transplantation surgery | 1 week after transplantation surgery
  number of subjects for which one or several dialysis session(s) is necessary until 1 week after transplantation surgery
Graft rejection rate 1 month after transplantation surgery | 1 month after transplantation surgery
  % of subjects with graft rejection until 1 month after transplantation surgery
Graft rejection rate 3 months after transplantation surgery | 3 months after transplantation surgery
  % of subjects with graft rejection until 3 months after transplantation surgery
Graft rejection rate 6 months after transplantation surgery | 6 months after transplantation surgery
  % of subjects with graft rejection until 6 months after transplantation surgery
Renal function 1 month after transplantation surgery | 1 month after transplantation surgery
  creatinine 1 month after transplantation surgery
Renal function 3 months after transplantation surgery | 3 months after transplantation surgery
  creatinine 3 months after transplantation surgery
Renal function 6 months after transplantation surgery | 6 months after transplantation surgery
  creatinine 6 months after transplantation surgery
Change in hemostasis parameters from before the desensitization protocol to after | the day of the first desensitization session (just before the session) and the day after the last desensitization session (up to 11 days)
  plasma level of fibrinogen clotting factors
Change in hemostasis parameters from before the desensitization protocol to after | the day of the first desensitization session (just before the session) and the day after the last desensitization session (up to 11 days)
  plasma level of factor XIII
Change in hemostasis parameters from before the desensitization protocol to after | the day of the first desensitization session (just before the session) and the day after the last desensitization session (up to 11 days)
  plasma level of thrombin-antithrombin complex
Change in hemostasis parameters from before the desensitization protocol to after | the day of the first desensitization session (just before the session) and the day after the last desensitization session (up to 11 days)
  plasma level of platelet secretion proteins (sCD40L, PF4)
Change in hemostasis parameters from before the desensitization protocol to after | the day of the first desensitization session (just before the session) and the day after the last desensitization session (up to 11 days)
  plasma level of ADAMTS13 metalloprotease
Change in hemostasis parameters from before the desensitization protocol to after | the day of the first desensitization session (just before the session) and the day after the last desensitization session (up to 11 days)
  Von Willebrand factor (cleaved form)
Change in hemostasis parameters from before the desensitization protocol to after | the day of the first desensitization session (just before the session) and the day after the last desensitization session (up to 11 days)
  blood level of platelet-monocyte complexes
Change in hemostasis parameters from before the desensitization protocol to after | the day of the first desensitization session (just before the session) and the day after the last desensitization session (up to 11 days)
  blood level of platelet-neutrophil polynuclear complexes
Change in hemostasis parameters from before the desensitization protocol to after | the day of the first desensitization session (just before the session) and the day after the last desensitization session (up to 11 days)
  endogenous thrombin potential
Change in hemostasis parameters from before the desensitization protocol to after | the day of the first desensitization session (just before the session) and the day after the last desensitization session (up to 11 days)
  peak thrombin

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud DEL BELLO, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital Toulouse (Hospital Rangueil), Toulouse, France

IPD SHARING:
Plan to Share IPD: No